CLINICAL TRIAL: NCT01806519
Title: A Motor Control Intervention of Patients With Forward Head Posture and Persistent Neck Pain - A Single System Experimental Design With 12 Month Follow-up
Brief Title: Motor_Control_Neck_SSED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luleå Tekniska Universitet (Other)
Responsible Party: Principal Investigator, Peter Michaelson, Senior lecturer, PhD., Luleå Tekniska Universitet
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: LTU_SG_5
Record Dates: First submitted 2013-03-04; First posted 2013-03-07 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Neck Pain; Forward Head Posture
Keywords: neck pain; motor control; intervention; forward head posture
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Motor control intervention of head posture — The tailored motor control intervention used for motor learning-procedure described by Fitts and Posner, further developed and adapted to rehabilitation of the spine by O´Sullivan.
  The stages involved in the process was the Cognitive stage, Associative stage and the Autonomous stage

SUMMARY:
Neck pain is a common problem in the western world. There is a group of people suffering from neck pain with a reduced ability to maintain an upright posture showing a forward head position and an altered muscle function.

The aim of the study was to evaluate a motor control intervention for patients with persistent neck pain and a forward head posture.

This pilot study used a Single System Experimental Design (SSED) with an A-B-A-design and multiple baselines.

The tailored motor control intervention addressed the faulty postural alignment and the deep muscles of the cervical spine.

ELIGIBILITY:
Inclusion Criteria:

* 20 - 50 years of age with pain originating from the neck for at least three months.
* A visual forward head posture.
* Less than105 points on the Örebro musculoskeletal pain screening questionnaire

Exclusion Criteria:

* neurological dysfunction.
* former cervical surgery or compression fracture of the spine
* no mental retardation
* no physiotherapy treatment during the last 6 months.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2009-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Head posture | Effect from baseline to 8 weeks and being maintained to 12 month
  The craniovertebral (CV) -angle was used to estimate the cervical curvature and head posture in relation to the thorax being measured with the Head Posture Spinal Curvature Instrument
Muscle function of the deep cervical flexors | Effect from baseline to 8 weeks and being maintained to 12 month
  The Cranio-Cervical Flexion Test (C-CFT) was used to assess the tonic holding abilities of the deep cervical muscles by using a Pressure biofeedback unit.

SECONDARY OUTCOMES:
Disability | Effect from baseline to 8 weeks and being maintained to 12 month
  The Neck Disability Index (NDI) is a self-reported questionnaire with 10 categories where each question estimates the current status, from no disability (0) to full disability within that category used to assess disability.
Pain intensity | Effect from baseline to 8 weeks and being maintained to 12 month
  The pain intensity was evaluated using the 100 mm Visual Analogue Scale (VAS) with the anchors "no pain" and "worst pain imaginable" that assessed the average pain intensity in the neck over the last seven days.

OTHER OUTCOMES:
Posture | Effect from baseline to 8 weeks and being maintained to 12 month
  The category Relation to Body Center (items Postural activity, Deviation in standing, Stability in stance and In sitting) and Relation to Ground (items Contact surface, Load, Stance on one leg) from the Body Awareness Scale (BAS) was used to measure the theoretical plumb line perpendicular to the body´s center to estimate the ability to maintain a neutral posture.

CONTACTS AND LOCATIONS:
Locations (1):
- OMT-kliniken, Luleå, Luleå, Sweden